CLINICAL TRIAL: NCT07096479
Title: A Real World Study on the Efficacy and Safety of Telpegfilgrastim Injection for Prophylaxis of Chemotherapy-Induced Neutropenia in Patients With Solid Tumor
Brief Title: Telpegfilgrastim Injection to Reduce the Risk of Neutropenia in Patients With Solid Tumor
Status: Recruiting | Type: Observational
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Lianxin Liu，PhD, chief physician, Anhui Provincial Hospital
Other Study IDs: PJ-B-05
Record Dates: First submitted 2024-08-05; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Chemotherapy-induced Neutropenia
Keywords: Drug Therapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Telpegfilgrastim Injection — Within 48 ± 12 hours after the end of each chemotherapy cycle, a single subcutaneous injection of a fixed dose of 2mg of Telpegfilgrastim is administered. Use once per chemotherapy cycle and enroll in 1-4 cycles based on the patient's actual condition.

SUMMARY:
The objective of this real world study is to confirm the efficacy and saftey of Telpegfilgrastim injection for the prevention of chemotherapy-induced Neutropenia in Patients With Malignant solid tumor.

DETAILED DESCRIPTION:
In recent years, the incidence rate of malignant tumors in China has increased year by year, and tumor treatment methods are also developing; However, various complications may still accompany the treatment of cancer patients, such as neutropenia, thrombocytopenia, nausea and vomiting. The treatment for neutropenia includes removal of the cause, supportive therapy, use of antibiotics, use of granulocyte colony-stimulating factor (G-CSF), oral medication, hematopoietic stem cell transplantation, hormone and immunotherapy, among which G-CSF is the most commonly used. At present, stratified management is recommended for chemotherapy-induced neutropenia, including primary prevention, secondary prevention, and treatment. For patients receiving high-risk chemotherapy regimens, prophylactic use of G-CSF is recommended, regardless of whether the treatment goal is to cure, prolong survival time, or improve disease-related symptoms. For patients receiving medium risk chemotherapy regimens, it is necessary to assess their own risk factors, such as patient age. If the patient meets any of the factors that increase the risk factor, it is recommended to use G-CSF preventively. The definition of secondary prevention of neutropenia is that if a patient develops FN or dose limiting neutropenia in the previous chemotherapy cycle, prophylactic use of G-CSF can be considered in the next chemotherapy cycle. For patients who have not received prophylactic use of G-CSF, a risk assessment of therapeutic use of rhG CSF should be conducted. If there are adverse factors, rhG CSF treatment should be considered.

Telpegfilgrastim is a Y-shaped polyethylene glycol (PEG) modified human granulocyte colony-stimulating factor (rhG-CSF) that has been approved by the NMPA for "reducing the incidence of infections manifested as febrile neutropenia in patients with non myeloid malignancies receiving bone marrow suppressive anticancer drugs that are prone to clinically significant febrile neutropenia. " Compared with the existing straight chain PEG rhG CSF in clinical practice, the Y-shaped branch structure of Telpegfilgrastim affects the activity and metabolic rate of the drug to a certain extent. While prolonging the half-life of the drug, the dosage is also significantly lower than that of long-acting products already on the market. It can be administered preventively after chemotherapy, maintaining the effective blood drug concentration throughout the entire cycle and effectively preventing the occurrence of neutropenia. Due to the reduction in medication dosage, the incidence of side effects such as skeletal and muscle pain is correspondingly reduced, resulting in better safety performance.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age ranging from 18 to 70 years old (excluding 70 years old);
2. body weight ≥45 kg;
3. Histologically or cytologically confirmed diagnosis of malignant solid tumor;
4. Solid tumor patients who receive a 3-week chemotherapy regimen have been evaluated as high-risk for FN or evaluated as having moderate risk for FN, but with an increased risk factor for neutropenia associated with the chemotherapy regimen;(The risk assessment of FN in tumor chemotherapy is based on " Chinese Society of Clinical Oncology (CSCO) guidelines for standardized management of tumor chemoradiotherapy related neutropenia(2021 edition)" and " Consensus on clinical diagnosis, treatment, and prevention of chemotherapy-induced neutropenia in China(2023 edition)";
5. Karnofsky Performance Scale(KPS) score≥70;
6. The total number of white blood cells and absolute value of neutrophils before chemotherapy should not be lower than normal values: WBC ≥ 3.5 × 109/L, ANC ≥ 1.5 × 109/L;
7. Subject has a life Expectation of at least 6 month；
8. Subjects voluntarily and strictly comply with the research protocol requirements and sign a written informed consent for.

Exclusion Criteria:

1. Received any other PEG-rhG-CSF within 4 weeks prior to participating in this study;
2. Patients receiving intermittent or continuous chemotherapy regimens such as albumin paclitaxel and capecitabine;
3. Previously or expected to receive extensive radiation therapy (>25% of total bone marrow);
4. Individuals with significant functional impairments in important organs such as the heart, lungs, liver, and kidneys:

   Liver function indicators (ALT, TBil)>2.5 ULN; Tumor patients with liver metastasis have liver function indicators (ALT,TBil)>5ULN; Hepatitis B virus infection, hepatitis C virus infection, or cirrhosis; Renal function Cr>1.5ULN;
5. Pregnant or breastfeeding woman ;
6. hypersensitive to rhG-CSF or other biological agents;
7. Investigators judged other situations that may affect the progress and results of clinical research.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Solid tumor patients who require chemotherapy (chemotherapy regimen for FN high-risk or FN medium risk accompanied by increased risk factors)
Sampling Method: Non-Probability Sample
Enrollment: 318 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2025-08-15 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
The incidence of grade ≥3 neutropenia during four chemotherapy cycles | At the end of each cycle (each cycle being 21 days)

CONTACTS AND LOCATIONS:
Locations (1):
- Anhui province hospital, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No